CLINICAL TRIAL: NCT02972801
Title: Testicular Tissue Cryopreservation for Fertility Preservation in Patients Facing Infertility-causing Diseases or Treatment Regimens
Brief Title: Testicular Tissue Cryopreservation for Fertility Preservation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Medical College of Wisconsin (Other); University of Chicago (Other); Helen DeVos Children's Hospital (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19020220
Record Dates: First submitted 2016-10-12; First posted 2016-11-23 (Estimated); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Autoimmune Disorders
Keywords: Spermatogonial stem cells; Testis; Fertility; Infertility; Oncofertility
MeSH Terms: conditions — Neoplasms; Autoimmune Diseases; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Testicular tissue biopsy (Experimental): Testicular biopsy
  Interventions: Procedure: Testicular biopsy

INTERVENTIONS:
Procedure: Testicular biopsy — Testicular biopsy is performed to obtain testicular tissue for cryopreservation

SUMMARY:
Testicular tissue cryopreservation is an experimental procedure where a young boy's testicular tissue is retrieved and frozen. This technique is reserved for young male patients who are not yet producing mature sperm, with the ultimate goal that their tissue may be used in the future to restore fertility when experimental techniques emerge from the research pipeline.

DETAILED DESCRIPTION:
Fertility status has an important impact on the post-treatment quality of life for cancer survivors and other patients that receive gonadotoxic therapies (e.g., prior to bone marrow transplantation). Semen cryopreservation is an established fertility preserving therapy, but is not accessible or appropriate for all men. Currently there are no therapies to preserve the future fertility of preadolescent boys. However, new reproductive therapies are under development and may one day offer "fertile hope" to those survivors that do not currently have access to fertility preserving therapies. Clinical management of fertility threatening diseases and treatments must have foresight of the gonadotoxic side effects and the potential for infertility. When no established fertility sparing options are available, it is reasonable to offer harvesting and cryopreservation of testicular tissue as a possible means of fertility preservation.

This study will harvest testicular tissue from eligible patients. Separate portions of the harvested tissue and/or cells will be 1) designated for research and 2) cryopreserved and maintained for participating patients as a resource for future elective procedures to attempt fertility restoration.

ELIGIBILITY:
Inclusion Criteria:

* Be male at any age.
* Be scheduled to undergo surgery, chemotherapy, drug treatment and/or radiation for the treatment or prevention of a medical condition or malignancy with risk of causing permanent and complete loss of subsequent testicular function.
* Or, have a medical condition or malignancy that requires removal of all or part of one or both testicles.
* Have newly diagnosed or recurrent disease. Those who were not enrolled at the time of initial diagnosis (i.e., patients with recurrent disease) are eligible if they have not previously received therapy that is viewed as likely to result in complete and permanent loss of testicular function.
* Have two testicles if undergoing elective removal of all or part of a testicle for fertility preservation only. Note: removal of both testicles will limit fertility preservation options.
* Sign an approved informed consent and authorization permitting the release of personal health information. The patient and/or the patient's legally authorized guardian must acknowledge in writing that consent for specimen collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and
* Consent for serum screening tests for infectious diseases [HIV-1, HIV-2, Hepatitis B, Hepatitis C], to be performed at the time of testicular tissue harvesting.
* Undergo a full history and physical examination and obtain standard pre-operative clearance (based on the most recent ACC/AHA Guideline for Perioperative Cardiovascular Evaluation for Noncardiac Surgery) as determined by their primary surgeon.
* Participating in long term follow-up is a requirement of the protocol.

Exclusion Criteria:

* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.
* Diagnosed with an underlying medical condition that significantly increases their risk of complications from anesthesia and surgery.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-01-06 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Presence of spermatogonial stem cells in the testicular tissue as determined by histology. | 5 years
  A segment of testicular specimen (~5%) will be removed and assessed for presence of spermatogonial stem cells by immunofluorescence and hematoxylin staining

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish individual participant data. The investigators will also report each individual participants data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: THe investigators will share IPD with the patient (and only the patient) within one year of enrollment. The investigators share study protocol and ICF with collaborating sites upon request. De-identified IDP is shared with collaborating sites annually.
Access Criteria: De-identified research data will be shared with collaborators via e-mail, and with the broader scientific community via publication and presentations at national/international meetings.